CLINICAL TRIAL: NCT05185973
Title: A Double Blinded Randomized Controlled, Community-based Trial in Rural Lao PDR to Determine the Positive Effects of "For Baby" Supplementation on Young Children's Physical Growth and a Reduction of Diarrhea Episodes
Brief Title: Effects of "For-Baby" Supplementation on Young Children's Physical Growth and Diarrhea Episodes
Acronym: LaoBiome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lao Tropical and Public Health Institute (Other Government)
Collaborators: Institut Pasteur du Laos (Unknown); Seoul National University (Other)
Responsible Party: Principal Investigator, Somphou SAYASONE, Head of Department, Lao Tropical and Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAO TROPICAL AND PUBLIC HEALTH
Record Dates: First submitted 2021-11-18; First posted 2022-01-11 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Children; Malnutrition
Keywords: Malnutrition; Nutrient supplementation; For-baby; Lao PDR
MeSH Terms: conditions — Malnutrition | interventions — Powders

STUDY DESIGN:
Intervention Model Description: The LaoBiome Study is a community-based double blinded randomized controlled trial. Approximately 1,200 infants and young children 6-23 months of age will be enrolled, and individually-randomized to one of two intervention groups of 600 children: 1) daily administration of For-Baby supplement (Intervention Group); 2) daily administration of micronutrient Placebo (Control Group). In both groups, children will remain under observation and receive their assigned supplements for a period of 12 months.
Who Masked: Participant, Investigator
Masking Description: The randomization scheme will be generated by an independent Statistician using a computer-generated block randomization scheme, with randomly selected block lengths of 4. Each of the two study arms will be identified by a unique 1-digit code (1, 2). The Institut Pasteur du Laos (IPL) member, unaffiliated with the study, will be responsible for assigning each of the two study codes to an intervention product and communicating this information directly to the product manufacturers. The identity of the treatment codes is stored in sealed envelopes held by the co-principal investigators (PIs) and the statistician. The envelopes will be opened only after statistical analyses of primary outcomes are completed and consensus on the interpretation of results is reached, unless required by one of the IRBs or the Project Steering Committee.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "For-Baby powder" supplement (Experimental): For-baby supplements provided as powder containing dry yeast powder, biovita mixed probiotics, synergy probiotics and other nutrients such as glucose, xylitol, chocolate powder, chocolate flavor powder, organic galactose oligosaccharide, chicory extract powder, vegetable Cream substitute, silicon dioxide, milk flavor powder, whole milk powder, zinc oxide, vitamin B12, vitamin B6, enzyme mixed preparation, vitamin C, organic alpha rice powder, folate 0.4mg, thiamine, leucin, isoleucin, valine, glutamine, and magnesium chloride.
  Interventions: Dietary Supplement: "For Baby "supplements provided as powder
- Micronutrient powder (Placebo Comparator): Micronutrient powder containing containing glucose 236.3mg, xylitol 150mg, chocolate powder 600mg, chocolate flavor powder 45mg, organic galactose oligosaccharide 60mg, chicory extract powder 60mg, vegetable Cream substitute 135mg, silicon dioxide 45mg, milk flavor powder 30mg, whole milk powder 75mg, zinc oxide 11.2mg, vitamin B12 2.6mg, vitamin B6 2mg, enzyme mixed preparation 2mg, vitamin C 1mg, organic alpha rice powder 1mg, folate 0.4mg, thiamine 0.5mg, and maltodextrin 1,541mg.
  Interventions: Dietary Supplement: Micronutrient powder provided as powder

INTERVENTIONS:
Dietary Supplement: "For Baby "supplements provided as powder — One sachet daily
  Arms: "For-Baby powder" supplement
Dietary Supplement: Micronutrient powder provided as powder — One sachet daily
  Arms: Micronutrient powder

SUMMARY:
The LaoBiome Study is a community-based, randomized, placebo-controlled trial with two study arms conducted in Lao People's Democratic Republic. This study aims at providing evidence on impact of For-baby powder supplement on child physical growth, diarrheal incidence, environmental enteric dysfunction, adherence to the intervention, and neuro-behavioural development of: 1) daily administration of For-Baby powder supplements (Intervention Group) and 2) daily administration of micronutrient powder (Placebo-Controlled Group).

DETAILED DESCRIPTION:
Probiotics are delivered as multiple micronutrient supplements in a powder package (For-Baby powder's sachet) and add into a single serving of clean water or breast milk and spoon feed the powder to the child 30 minutes before or after food consumption or add to semi-solid or mashed food such as mashed mango, banana and papaya, boiled pumpkin, and boiled egg after the food has been cooked and cooled sufficiently to be eaten (but within 30 minutes of preparation). Recent studies has shown that certain probiotics are extremely useful for the treatment of environmental enteropathy in malnourished children and has significant growth promoting effects. Nonetheless, new studies are needed to better understand the environmental enteropathy and its consequences.

This community-based, randomized, placebo-controlled trial with two groups will be conducted in the community of Luangprabang province in the northern part of Lao PDR.

The study team will enroll a total of 1,200 children, aged 6-23 months into the trial. The children will be randomly assigned one of two groups: 1) intervention group of daily For-Baby powder supplements and 2) control group of daily micronutrient powder supplements. After enrollment, the children will be under the observation for a total of 12 months (52 weeks). The monitored outcomes are the physical growth, diarrheal episodes, motor and intellectual development, gut microbiota and intestinal parasitic infections.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-23 months of age at enrollment,
* Acceptance of weekly home visits for growth surveillance,
* Planned residency within the study area for the duration of the study period (52 weeks),
* Signed informed consent from a parent or legal caregiver.

Exclusion Criteria:

* Weight-for-height z-score (WHZ) <-3SD with respect to World Health Organization 2006 standards;
* Presence of bipedal edema;
* Severe illness warranting hospital referral;
* Congenital abnormalities potentially interfering with growth;
* Chronic medical condition (e.g., malignancy) requiring frequent medical attention;
* Known human immunodeficiency virus (HIV) infection of index child or child's mother;
* Severe anemia (hemoglobin <70 g/L; based on testing at enrollment);
* Currently consuming MNP supplements;
* Current participation in any other clinical trial.

Criteria for discontinuation:

A subject can be discontinued from the study for the following reasons:

* Withdraws from the study (this can happen anytime as participation is voluntary and there are no further obligations).
* At the discretion of the principal investigator, if the participant is not compliant to the requirements of the protocol.
* Discontinued subjects will not be replaced. If, for any reason, a subject is discontinued from the study before the end of the evaluations, the safety procedures planned (AEs monitoring) will be conducted. Data obtained prior to subject's withdrawal will be included in analysis. Data of withdrawn patients are fully anonymized once analysis is completed.

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2023-02-19 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in length and length-for-age Z-score | 52 weeks
  Length of study children will be measured at the baseline, and follow-up surveys using seca baby's length measuring board.
Change in weight and weight-for-age Z-score, | 52 weeks
  Weight of study children will be measured at the baseline, and follow-up surveys, using seca baby's digital scale.
Change in mid-upper circumference | 52 weeks
  Mid- upper arm circumference will be measured the baseline, and follow-up surveys, using a mid upper arm circumference measuring tape.

SECONDARY OUTCOMES:
Incidence of diarrheal episodes | 52 weeks
  Report of diarrheal episodes will be recorded at the baseline and follow-up surveys
Number of children achieved the gross motor developmental milestones | 52 weeks
  Gross motor developmental milestones as recommended by the World Health Organization include: sitting without support, crawling, standing with assistance, walking with assistance, standing alone, walking alone
Number of children with improved gut microbiota profile | 52 weeks
  Gut microbiota will be assessed using microbiome analysis
Intestinal protozoa infection | 52 weeks
  Intestinal protozoan infections will be assessed by a modified formalin-ethyl acetate concentration technique
Helminth parasitic infection | 52 weeks
  Helminth parasitic infections will be assessed using duplicate Kato-Katz thick smears

CONTACTS AND LOCATIONS:
Overall Officials: Latsamy P Siengsounthone, MD, Study Director — Lao Tropical and Public Health Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schroder L, Kaiser S, Flemer B, Hamm J, Hinrichsen F, Bordoni D, Rosenstiel P, Sommer F. Nutritional Targeting of the Microbiome as Potential Therapy for Malnutrition and Chronic Inflammation. Nutrients. 2020 Oct 3;12(10):3032. doi: 10.3390/nu12103032. PMID 33022941
- [Background] Maldonado NC, Chiaraviglio J, Bru E, De Chazal L, Santos V, Nader-Macias MEF. Effect of Milk Fermented with Lactic Acid Bacteria on Diarrheal Incidence, Growth Performance and Microbiological and Blood Profiles of Newborn Dairy Calves. Probiotics Antimicrob Proteins. 2018 Dec;10(4):668-676. doi: 10.1007/s12602-017-9308-4. PMID 28770479
- [Background] Vadopalas L, Zokaityte E, Zavistanaviciute P, Gruzauskas R, Starkute V, Mockus E, Klementaviciute J, Ruzauskas M, Lele V, Cernauskas D, Klupsaite D, Dauksiene A, Sederevicius A, Badaras S, Bartkiene E. Supplement Based on Fermented Milk Permeate for Feeding Newborn Calves: Influence on Blood, Growth Performance, and Faecal Parameters, including Microbiota, Volatile Compounds, and Fatty and Organic Acid Profiles. Animals (Basel). 2021 Aug 30;11(9):2544. doi: 10.3390/ani11092544. PMID 34573514
- [Background] Barkhidarian B, Roldos L, Iskandar MM, Saedisomeolia A, Kubow S. Probiotic Supplementation and Micronutrient Status in Healthy Subjects: A Systematic Review of Clinical Trials. Nutrients. 2021 Aug 28;13(9):3001. doi: 10.3390/nu13093001. PMID 34578878
- [Background] Hajare ST. Effects of potential probiotic strains LBKV-3 on Immune Cells responses in Malnutrite children: a double-blind, randomized, Controlled trial. J Immunoassay Immunochem. 2021 Sep 3;42(5):453-466. doi: 10.1080/15321819.2021.1895217. Epub 2021 Mar 22. PMID 33750266
- See also: All references are published online in the peer reviewed journals — https://pubmed.ncbi.nlm.nih.gov